CLINICAL TRIAL: NCT01950065
Title: Effectiveness and Safety Study of the Iovera Device for the Temporary Reduction in the Appearance of Forehead Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYO-0806
Record Dates: First submitted 2013-09-17; First posted 2013-09-25 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Forehead Wrinkles

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Immediate Treatment with iovera (Experimental): Immediate treatment with iovera
  Interventions: Device: iovera
- Delayed Treatment with iovera (Active Comparator): Delayed Treatment with iovera
  Interventions: Device: iovera

INTERVENTIONS:
Device: iovera

SUMMARY:
Evaluate the effectiveness and safety of the iovera device for the temporary reduction in the appearance of forehead wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Subject has a forehead wrinkle rating by the Investigator/designee of at least "2" in full contraction on the 5-point Wrinkle Scale (5WS) as rated by the study Investigator, which, upon physical manipulation/separation of the skin, demonstrates a reduction in wrinkle severity
* Subject has a glabella wrinkle rating by the Investigator/designee of at least "1" in full contraction on the 5-point Glabella Scale (5GS)
* Subject has at least a 2 point difference between resting and dynamic forehead wrinkle scores using the 5-point Wrinkle Scale (5WS) as rated by the Investigator/designee
* Subject has Fitzpatrick Skin Type I, II, III, or IV (see Error! Reference source not found.)
* Subject understands and commits to comply with study requirements
* Subject is in good general health and free of any condition that could impair either complete study participation or evaluation of forehead wrinkle rating
* Subject is willing and able to give written informed consent

Exclusion Criteria:

* Subject has a clotting disorder or coagulopathy that requires regular use of an anticoagulant and/or antiplatelet therapy (e.g., warfarin, clopidogrel, etc.)
* Subject has used aspirin or any non-steroidal anti-inflammatory drugs (NSAIDs) within seven (7) days prior to screening or use of the device
* Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites
* Subject has undergone another surgical cosmetic procedure or botulinum toxin injection at or above the level of the zygoma (cheekbones) within the past six (6) months prior to screening
* Subject has a resting wrinkle score of "3" or higher on the 5WS as rated by the study Investigator
* Subject actively elevates forehead during rest
* Subject has been treated with any fillers listed in Error! Reference source not found. in the temple or forehead area in the time intervals specified prior to screening
* Subject has any of the following conditions:

  * Dermatochalasis with <2mm lid margin when looking straight ahead
  * Excessive skin laxity/skin aging
  * Asymmetry in the upper face
  * History of facial nerve palsy
  * Eyebrow or eyelid ptosis
  * History of neuromuscular disorder
  * Chronic dry eye symptoms
  * Allergy or intolerance to local anesthetic agents (e.g., Lidocaine)
  * Use of narcotic medications for a chronic pain condition
  * Other clinically significant local skin condition (e.g., skin infection) at target treatment site
  * Any physical or psychiatric condition that in the Investigator's opinion would prevent treatment or adequate study participation
  * Chronic medical condition that in the Investigator's opinion would affect study participation (such as diabetes, hepatitis, HIV, etc.)
  * Known diagnosis of cryoglobulinemia, paroxysmal cold hemoglobinuria, or cold urticaria
  * Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the Investigator
* Fitzpatrick Skin Type V or VI (see Table 3)
* Subject currently enrolled in an investigational drug, biologic or device study that could affect the safety or effectiveness of wrinkle treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Improvement on the 5-point Wrinkle Scale | 30 Days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Roseville Facial Plastic Surgery, Roseville, California
  - DeNova Research, Chicago, Illinois
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - Laser & Skin Surgery Center of NY, New York, New York
  - Nashville Center for Laser and Facial Surgery, Nashville, Tennessee
  - Dallas Plastic Surgery Institute, Dallas, Texas